CLINICAL TRIAL: NCT01432899
Title: Characteristics and Mechanism of Childhood-Onset Hemidystonia
Brief Title: Studying Childhood-Onset Hemidystonia
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Other Study IDs: 110246; 11-CC-0246
Record Dates: First submitted 2011-09-10; First posted 2011-09-13 (Estimated); Last update posted 2018-12-24 (Actual); Status verified 2018-12-20

CONDITIONS: Dystonia; Cerebral Palsy
Keywords: Neurophysiology; Hemidystonia; Childhood-onset; Motion Analysis; Neuroimaging; Childhood Onset Hemidystonia; Healthy Volunteer; HV
MeSH Terms: conditions — Dystonia; Cerebral Palsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

SUMMARY:
Background:

- Childhood-onset dystonia is caused by a brain injury. It causes muscle contractions and twisting movements that the person with dystonia cannot control. The term hemidystonia is used when only one side of the body is affected. When dystonia starts during childhood, the brain and nerves may not develop normally. People with hemidystonia can become disabled because of the unwanted postures and twisting that dystonia causes. More research is needed to determine how dystonia affects brain development.

Objectives:

- To study brain function in people with hemidystonia.

Eligibility:

* Individuals between 18 and 40 years of age who developed hemidystonia before age 13. Only one wrist may be affected by hemidystonia, and participants must have at least some movement in that wrist.
* Healthy volunteers at least 18 years of age.

Design:

* This study requires five visits to the NIH Clinical Center: a screening visit and four study visits. Each visit will last up to 3 hours. Visits will be scheduled about once a week. The study procedures may be done in any order.
* Participants will be screened with a physical exam and medical history.
* Participants will have the following tests:
* Brain magnetic resonance imaging scan. During the scan, participants will be asked to move their hand at the wrist when they hear a tone.
* Motor tests of arm movement, balance, and walking. These tests may also examine nerve development and muscle tone.
* Two transcranial magnetic stimulation sessions to study the electrical activity of the muscles and brain. These sessions may also involve sensory tests. Participants will have hearing tests before the first session and after the second session.
* No treatment for hemidystonia will be provided as part of this study.

DETAILED DESCRIPTION:
Objective

In childhood-onset hemidystonia, motor and sensory abnormalities pose a great challenge to voluntary movement. In an effort to inform future methods of treatment of this disorder, this study seeks to (1) characterize involuntary muscle activity, (2) explore neurophysiologic mechanisms of involuntary muscle activity, (3) characterize abnormalities of sensation, (4) assess performance on two sensorimotor tasks (voluntary postural control, and a reach-to-grasp arm movement), and (5) explore brain abnormalities using imaging in childhood-onset hemidystonia.

Study Population

The dystonia group will consist of 40 individuals (age 7-40 years) with childhood-onset hemidystonia. The control group will consist of 40 individuals within the same age range with no neurological disorders.

Design

This is a cross-sectional study, in which multiple assessments will be performed over a short period. Results in the dystonia group will be compared to results in the control group. Due to the laterality of brain injury in hemidystonia, outcomes from both arms and cortical hemispheres will be compared to each other. Outcomes within the dystonia group will be correlated with validated dystonia rating scales as well as with the age at the time of injury.

Outcome Measures

In Objective 1, we will analyze the timing of involuntary electromyographic (EMG) activity and kinematics triggered in the dystonic arm during various tasks. In Objective 2, we will investigate various types of intracortical inhibition (short intracortical inhibition, long intracortical inhibition, contralateral silent period, and ipsilateral silent period) and intracortical facilitation in motor cortical regions controlling the dystonic wrist flexor during voluntary contraction of the wrist extensor using transcranial magnetic stimulation (TMS). In addition, we will perform a coherence analysis between EMG activity in the wrist flexor and extensor muscles and between electroencephalographic (EEG) activity in the primary motor cortex and the contralateral wrist muscles. In Objective 3, we will test tactile sense (spatial and temporal), vibration sense, and stereognosis of the hand. In Objective 4, we will analyze seated limits of stability (voluntary postural control), and the timing and amplitude of EMG activity and kinematics in the arm during a reaching and grasping arm movement. In Objective 5, we will obtain brain scans with structural magnetic resonance imaging (MRI), diffusion tensor imaging (DTI), resting state functional connectivity MRI, and functional MRI during a simple task.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age 7 40 years, inclusive
* Good general health, with enough energy to carry out the assessments
* Ability to understand and comply with instructions. Adults must be able to provide their own consent.
* Passive motion of at least 15 degrees extension and 15 degrees flexion from neutral of both wrist joints
* Agreement to not drink caffeine or alcohol for 24 hours before each study session because both agents can modify brain activity and may confound outcome measures.

Additional inclusion criteria for individuals with dystonia:

- Childhood-onset (before 13 years of age) hemidystonia in one wrist. Diagnosis of dystonia will be made based on the Hypertonia Assessment Tool (HAT)

EXCLUSION CRITERIA:

Healthy Volunteers:

-Presence of any neurological disorders

Individuals with Dystonia:

* Botulinum toxin injection in the flexor carpi radialis and extensor carpi radialis in the last 6 months
* Concurrent use of medicines for muscle tone (e.g., baclofen, trihexyphenedyl, dantrolene sodium, tizanidine, or carbidopa/levodopa). If patients are taking these medications daily, the treating physician will be contacted by the MAI to determine if it is acceptable for the subject to temporarily discontinue the medication(s). If the risk of weaning, or stopping the medication is deemed harmless, the MAI and/or treating physician will determine a schedule to wean, or stop the medication. The goal is for the subject to be off medication(s) for 24 hours prior to participating in testing for this study. For these subjects, there will be at least 4 days between scheduled research visits to avoid a prolonged time off medication(s).

Additional exclusion criteria for TMS:

* Seizure in the last 2 years
* Concurrent use of anti-seizure medication
* Hearing loss
* Cardiac pacemakers, implanted medication pumps, intracardiac lines, or acute, unstable cardiac disease, with intracranial implants (e.g. aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or any other metal object within or near the head, excluding the mouth that cannot be safely removed.

Additional exclusion criteria for MRI:

* Inability to lie flat on the back for up to 1 hour
* Uncontrolled movements of the head when lying supine as determined by the MAI
* Discomfort being in small spaces for up to 1 hour
* Cardiac pacemakers, implanted medication pumps, intracardiac lines, or acute, unstable cardiac disease, with intracranial implants (e.g. aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or any other metal object within or near the head, excluding the mouth that cannot be safely removed.
* Pregnancy: For any female of childbearing potential, a pregnancy test will be done. Childbearing potential will be determined during the history and physical.

Ages: 7 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 21 (Actual)
Dates: Start 2011-09-10; Study Completion 2018-12-20

PRIMARY OUTCOMES:
Sum of wrist, elbow, and shoulder excursion
Difference between the peak-to-peak amplitude of MEP due to the TS and the CS for SICI.
Performance accuracy on sterognosis.
Maximum excursion and Time to largest hand aperture

SECONDARY OUTCOMES:
This protocol has 5 Objectives, each with its own primary and secondary objectives. They are too numerous to list.

CONTACTS AND LOCATIONS:
Overall Officials: Diane L Damiano, Ph.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Abbruzzese G, Berardelli A. Sensorimotor integration in movement disorders. Mov Disord. 2003 Mar;18(3):231-240. doi: 10.1002/mds.10327. PMID 12621626
- [Background] Aertsen AM, Gerstein GL, Habib MK, Palm G. Dynamics of neuronal firing correlation: modulation of "effective connectivity". J Neurophysiol. 1989 May;61(5):900-17. doi: 10.1152/jn.1989.61.5.900. PMID 2723733
- [Background] Albanese A, Barnes MP, Bhatia KP, Fernandez-Alvarez E, Filippini G, Gasser T, Krauss JK, Newton A, Rektor I, Savoiardo M, Valls-Sole J. A systematic review on the diagnosis and treatment of primary (idiopathic) dystonia and dystonia plus syndromes: report of an EFNS/MDS-ES Task Force. Eur J Neurol. 2006 May;13(5):433-44. doi: 10.1111/j.1468-1331.2006.01537.x. PMID 16722965
- [Derived] de Campos AC, Kukke SN, Hallett M, Alter KE, Damiano DL. Characteristics of bilateral hand function in individuals with unilateral dystonia due to perinatal stroke: sensory and motor aspects. J Child Neurol. 2014 May;29(5):623-32. doi: 10.1177/0883073813512523. Epub 2014 Jan 5. PMID 24396131